

### TRIAL STATISTICAL ANALYSIS PLAN

c28702727-01

**BI Trial No.:** 1402-0010

**Title:** Relative bioavailability and food effect of a single dose of different

solid formulations of BI 1358894 compared to a single dose of the

reference tablet formulation of BI 1358894 following oral administration under fed and fasted conditions in healthy male subjects (an open-label, single-dose, randomised, incomplete

blocks crossover design study)

Including Protocol Amendment 2 [c26426667-03]

Investigational

**Product:** 

BI 1358894

Responsible trial statistician:

Phone: Fax:

Date of statistical analysis plan:

06 AUG 2019 SIGNED

anarysis pian.

Version: Final


**Proprietary confidential information** 

© 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

TSAP for BI Trial No: 1402-0010 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 1 | TARLE | OF CONTENTS |
|----|-------|-------------|
| 1. | | |

| TITLE | PAGE | 1 |
|------------|----------------------------------------------|---|
| 1. | TABLE OF CONTENTS | 2 |
| LIST O | F TABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | 5 |
| 3. | INTRODUCTION | 7 |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | 8 |
| 5. | ENDPOINTS | 9 |
| <b>5.1</b> | PRIMARY ENDPOINTS | 9 |
| <b>5.2</b> | SECONDARY ENDPOINTS | 9 |
| 5.2.1 | Key secondary endpoints | 9 |
| 5.2.2 | Secondary endpoints | |

| <b>6.</b> | GENERAL ANALYSIS DEFINITIONS | 11 |
|---|---|---|
| 6.1 | TREATMENTS | |
| 6.2 | IMPORTANT PROTOCOL DEVIATIONS | 13 |
| 6.3 | SUBJECT SETS ANALYSED. | |
| 6.5 | POOLING OF CENTRES | 15 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | 15 |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | |
| 7. | PLANNED ANALYSIS | 17 |
| <b>7.1</b> | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION | 18 |
| 7.3 | TREATMENT COMPLIANCE | 18 |
| 7.4 | PRIMARY ENDPOINTS | |
| 7.4.1 | Primary analysis of the primary endpoints | |
| 7.4.2 | Sensitivity analysis, subgroup analysis, exploratory analysis of the primary endpoints | |
| 7.5 | SECONDARY ENDPOINTS | |
| 7.5.1 | Key secondary endpoints | |
| 7.5.2 | Secondary endpoints | |

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1402-0010 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 7.7 | EXTENT OF EXPOSURE | 20 |
|--------------|--------------------|----|
| <b>7.8</b> | SAFETY ANALYSIS | 20 |
| <b>7.8.1</b> | Adverse Events | 20 |
| 7.8.2 | Laboratory data | 22 |
| 7.8.3 | Vital signs | |
| 7.8.4 | ECG. | |
| 7.8.5 | Others | 22 |
| 8. | REFERENCES | 24 |
| 10. | HISTORY TABLE | 26 |

Boehringer Ingelheim
TSAP for BI Trial No: 1402-0010
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# **LIST OF TABLES**

| Table 6.1: 1 | Dosage and treatment schedule of BI 1358894 | 11 |
|---|---|---|
| Table 6.1: 2 | Analysis phases for statistical analysis of AEs, safety laboratory and vital | |
| | signs | 12 |
| Table 6.2: 1 | Handling of IPDs | |
| Table 6.3: 1 | Subject sets analyzed | 15 |
| Table 10: 1 | History table | 26 |

TSAP for BI Trial No: 1402-0010 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### LIST OF ABBREVIATIONS 2.

| Term | Definition / description |
|---|---|
| ADME | Absorption, Distribution, Metabolism and Excretion |
| AE | Adverse Event |
| AESI | Adverse event of special interest |
| ALT | Alanine aminotransferase |
| ANOVA | Analysis of variance |
| AST | Aspartate aminotransferase |
| AUC <sub>0-72</sub> | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 72 h |
| $\mathrm{AUC}_{0	ext{-tz}}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point |
| $\mathrm{AUC}_{0\text{-}\infty}$ | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity |
| BI | Boehringer Ingelheim |
| BP | Blood pressure |
| $C_{\text{max}}$ | Maximum measured concentration of the analyte in plasma |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| CV | Arithmetic coefficient of variation |
| C-SSRS | Columbia Suicidal Severity Rating scale |
| ECG | Electrocardiogram |
| gCV | geometric coefficient of variation |
| gMean | Geometric mean |
| ICH | International Conference On Harmonisation |
| IPD | Important protocol deviations |
| IQRMP | Integrated quality and risk management plan |
| MedDRA | Medical Dictionary For Regulatory Activities |
| PK | Pharmacokinetics |
| PKS | Pharmacokinetic parameter set |
| PR | Pulse rate |
| RAGe | Report appendix generator |

Boehringer Ingelheim
TSAP for BI Trial No: 1402-0010 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|------|---------------------------------|
| SAE | Serious adverse event |
| SD | Standard Deviation |
| SOC | System Organ Class |
| TS | Treated set |
| TSAP | Trial Statistical Analysis Plan |
| ULN | Upper limit of normal range |

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 3. INTRODUCTION

As per ICH E9 (1) the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the revised CTP, and to include detailed procedures for executing the statistical analysis of the primary variables and other data.

This TSAP assumes familiarity with the CTP and its amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the revised CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation.

Study data will be stored in a trial database within Medidata Rave system.

The statistical analyses will be performed within the validated working environment CARE, including SAS<sup>TM</sup> (current Version 9.4, by SAS Institute Inc., Cary, NC, USA), and a number of SAS<sup>TM</sup>-based tools (e.g., macros for the analyses of AE data or laboratory data; Report Appendix Generator system (RAGe) for compilation/formatting of the CTR appendices).

PK parameters will be calculated using Phoenix WinNonlin<sup>TM</sup> software (version Phoenix 6.3, Certara USA Inc., Princeton, NJ, USA).

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

The CTP states in Section 7.3.4 that AEs occurring after the residual effect period but prior to next intake or end of trial termination date will be assigned to "follow-up". As a more conservative approach, all AEs occurring after intake of trial medication and prior to next intake or end of trial termination date will be assigned to the on-treatment period of the respective trial medication. I.e., no follow-up phases will be defined in this trial, cf. Table 6.1: 2.

All other analyses described in this TSAP are in accordance with the statistical methods described in the revised CTP.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 5. ENDPOINTS

### 5.1 PRIMARY ENDPOINTS

Primary endpoints are PK endpoints of BI 1358894, as defined in Section 2.1.2 of the CTP:

- $C_{max}$  (maximum measured concentration of the analyte in plasma)
- $AUC_{0-tz}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point)

### 5.2 SECONDARY ENDPOINTS

# 5.2.1 Key secondary endpoints

Not applicable.

### 5.2.2 Secondary endpoints

Secondary endpoints are PK endpoints of BI 1358894, as defined in Section 2.1.3 of the CTP:

- $AUC_{0-\infty}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity)
- $AUC_{0-72}$  (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to 72 h)

TSAP for BI Trial No: 1402-0010 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 6. GENERAL ANALYSIS DEFINITIONS

### 6.1 TREATMENTS

For basic study information on treatments to be administered, assignment of treatment groups, and selection of doses, cf. Section 4 of the CTP.

Each subject is planned to be treated in three subsequent treatment periods, with one single dose in each treatment period. Subjects will receive three out of the five BI 1358894 treatments described in Table 6.1: 1.

Table 6.1: 1 Dosage and treatment schedule of BI 1358894

| Product | Treatment | Formulation | Unit<br>strength | Dosage | Total dose |
|---|---|---|---|---|---|
| TF2 | В | Tablet | 50 mg | 2 tablets (50 mg), single dose, fed | 100 mg |
| | C | Tablet | 50 mg | 2 tablets (50 mg), single dose, fasted | 100 mg |
| TF2 | D | Tablet | 50 mg | 2 tablets (50 mg), single dose, fed | 100 mg |
| | E | Tablet | 50 mg | 2 tablets (50 mg), single dose, fasted | 100 mg |
| TF1 | A | Tablet | 100 mg | 1 tablet (100 mg), single dose, fed | 100 mg |

Each subject is planned to be randomly allocated to one of twelve treatment sequences.

<u>Table 6.1: 2</u> shows definitions of analysis phases within each subject for statistical analyses of AEs, safety laboratory and vital signs.

Table 6.1: 2 Analysis phases for statistical analysis of AEs, safety laboratory and vital signs

| phase | Label | | Start | End |
|---|---|---|---|---|
| Screening | Screeni | ng | Date of informed consent | Date/time of first administration of BI 1358894 |
| On treatment | TF2 TF2 fed, TF2 fas or TF1 fed respective | - | Date/time of administration of<br>the respective formulation of<br>BI 1358894 | Date/time of administration of study drug in the next treatment period or 0:00 AM on day after subject's end of study participation date, whatever comes first |

AE displays in CTR Section 15.3, Appendix 16.1.13.1.8.2 and Appendix 16.1.13.1.8.3 will present results for the on-treatment phase only.

In AE tables in CTR Section 15.3 (but not in Appendix 16.1.13.1.8.2 and Appendix 16.1.13.1.8.3 AE tables), the following total will be provided in addition:

• "Total on-trt", defined as the total over all on-treatment phases

CTR Appendix 16.1.13.1.8.1 displays will present results for the screening and on-treatment phases.

Additionally to the total defined above, the following total will be provided in AE tables in CTR Section 16.1.13.1.8.1:

• "Total", defined as the total over all study phases (screening + on-treatment)

Statistical analyses of safety laboratory tests and vital signs will be conducted by treatment period , with clear differentiation between baseline (cf. Section 6.7) and on-treatment measurements (as defined in Table 6.1: 2).

More details on the technical implementation of these analyses are provided in the ADS Plan of this TSAP.

TSAP for BI Trial No: 1402-0010 Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 6.2 IMPORTANT PROTOCOL DEVIATIONS

Consistency check listings (for identification of deviations from time windows) and a list of protocol deviations (e.g. deviations in drug administration, in blood sampling times, etc.) will be provided to be discussed at the Report Planning Meeting. At this meeting, it will be decided whether a discrepant data value can be used in analyses or whether it must be corrected in the clinical database. Each protocol deviation must be assessed to determine whether it is an IPD. For definition of IPDs, and for the process of identification of these, refer to the BI reference document "Identify and Manage Important Protocol Deviations (IPD)" (2).

If any IPDs are identified, they are to be summarised into categories and will be captured in the decision log. Categories which are considered to be IPDs in this trial are defined in the integrated quality and risk management plan (IQRMP). If the data show other IPDs, the definition in the IQRMP will be supplemented accordingly by the time of the Report Planning Meeting.

IPDs will be summarized and listed. Table 6.2: 1 below specifies which kind of IPDs could potentially lead to exclusion from which analysis set. The decision on exclusion of subjects from analysis sets will be made at the latest at the Report Planning Meeting, after discussion of exceptional cases and implications for analyses. If the data show other IPDs, this table will be supplemented accordingly by the time of the Report Planning Meeting.

TSAP for BI Trial No: 1402-0010 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 6.2: 1 Handling of IPDs

| IPD code | IPD Category & Brief Description | Excluded from which analysis set |
|---|---|---|
| A1 | Inclusion Criteria Not Met | PKS |
| A2 | Exclusion Criteria Violated | PKS |
| B1 | Informed consent not available/not done | TS, PKS |
| B2 | Informed consent too late | None |
| C1 | Incorrect trial medication taken | PKS |
| C2 | Randomization not followed | PKS |
| C3 | Non-compliance | PKS |
| C4 | Incorrect intake of trial medication | PKS |
| C5 | Improper washout between treatments | PKS |
| D1 | Prohibited medication use | PKS |
| D2 | Mandatory medication not taken | PKS |
| D3 | Improper washout of concomitant medication | PKS |
| E1 | Certain violations of procedures used to measure primary or secondary data | PKS |
| F1 | Certain violations of time schedule used to measure primary or secondary data | PKS |
| G1 | Incorrect intake of meal | PKS |
| G2 | C-SSRS not conducted at discharge and EOT | None |

### 6.3 SUBJECT SETS ANALYSED

Subject sets will be used as defined in the CTP, Section 7.3.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 6.3: 1 Subject sets analyzed

| | Subject set | |
|----------------------------------------|-------------|-----|
| Class of endpoint | TS | PKS |
| Primary PK endpoints | | X |
| Secondary PK endpoints | | X |
| Safety parameters & treatment exposure | X | |
| Demographic/baseline endpoints | X | |

### 6.5 POOLING OF CENTRES

This section is not applicable, because the study was performed in only one centre.

# 6.6 HANDLING OF MISSING DATA AND OUTLIERS

Data of screened subjects who were withdrawn from the trial prior to first administration of any study drug will not be reported in the CTR.

Data of subjects who failed to complete all periods of the study (dropouts or withdrawals) will be reported in the CTR as far as their data are available. All withdrawals will be documented and the reason for withdrawal reported in the CTR.

**CTP**: *It is not planned to impute missing values for safety parameters.* 

One exception where imputation might be necessary for safety evaluation are AE dates. Missing or incomplete AE dates are imputed according to BI standards (3).

Missing data and outliers of PK data are handled according to BI standards (4). **CTP**: *PK parameters that cannot be reasonably calculated based on the available drug concentration-time data will not be imputed.* 

### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

A separate baseline is defined for each study treatment:

- Baseline for the treatment in the first treatment period is defined as the last available off-treatment value before administration of the respective formulation of BI 1358894.
- Baseline for the treatment in the second and third treatment periods is defined as the last available pre-dose value measured on or after Day 14 of the preceding visit.

Time windows are defined in Section 6.1 of the CTP. Adherence to time windows will be checked at the Report Planning Meeting.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### 7. PLANNED ANALYSIS

The format of the listings and tables will follow the BI guideline "Reporting of clinical trials and project summaries" (5).

The individual values of all subjects will be listed. Listings will be sorted by treatment sequence, subject number and visit (if visit is applicable in the respective listing). AE listings will be sorted by assigned treatment (see Section 7.8.1 below for details). The listings will be contained in Appendix 16.2 (SDL) of the CTR.

The following standard descriptive statistical parameters will be displayed in summary tables of continuous variables:

N number of non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For plasma concentrations as well as for all PK parameters the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

For PK parameters the following descriptive statistics will additionally be calculated:

P10 10<sup>th</sup> percentile Q1 1<sup>st</sup> quartile Q3 3<sup>rd</sup> quartile P90 90<sup>th</sup> percentile

The data format for descriptive statistics of plasma concentrations will be identical with the data format of the respective concentrations. The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group. Percentages will be rounded to one decimal place. The category missing will be displayed if and only if there actually are missing values. Percentages will be based on all subjects in the respective subject set whether they have non-missing values or not.

TSAP for BI Trial No: 1402-0010 Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the CTR.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Concomitant diseases will be coded according to the most recent version of MedDRA. Concomitant medication will be coded according to the most recent version of the World Health Organisation – Drug Dictionary. Concomitant non-drug therapies will be coded according to the most recent version of MedDRA.

Only descriptive statistics are planned for this section of the CTR.

#### 7.3 TREATMENT COMPLIANCE

Treatment compliance will not be analyzed as a specific endpoint. Any deviations from complete intake will be addressed in the Report Planning Meeting (cf. Section 6.2) and described in the CTR.

#### 7.4 PRIMARY ENDPOINTS

#### 7.4.1 Primary analysis of the primary endpoints

Primary analysis of the primary endpoints will be performed as defined in Sections 7.3.1 of the CTP.

The statistical model for the primary analysis defined in the CTP is an analysis of variance (ANOVA) model on the logarithmic scale including "treatment", "period" and "sequence" as fixed effects and "subjects within sequences" as random effect. Relative bioavailability of the study treatments will be estimated by the ratios of the geometric means

- C/A, i.e. TF2 fas/TF1 fed
- E/A, i.e.TF2 fas/ TF1 fed, i.e.
- B/C, i.e. TF2 fed/TF2 fas
- D/E, i.e. TF2 fed/TF2 fas

of the primary endpoints.

### Exclusion of PK parameters

The ADS ADPP contains column variables APEXC and APEXCO indicating inclusion/exclusion (APEXC) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS are based on PK parameter values which are not flagged for exclusion, i.e. with APEXC equal to "Included".

### Exclusion of plasma concentrations

The ADS ADPC (PK concentrations per time-point or per time-interval) contains column variables ACEXC or ACEXCO indicating inclusion/exclusion (ACEXC) of a concentration

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to "ALL CALC", the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to "DESC STATS" the value will be excluded from descriptive evaluations per planned time point/time interval. If ACEXCO contains the addition "TIME VIOLATION" or "TIME DEVIATION", the value can be used for further analyses based on actual times. If ACEXCO is set to "HALF LIFE", the value will be excluded from half-life calculation only; the value is included for all other analyses. Excluded concentration itself will be listed in the CTR associated with an appropriate flag.

Further details are given in "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (4) and "Description of Analytical Transfer Files and PK/PD Data Files" (6).

# 7.4.2 Sensitivity analysis, subgroup analysis, exploratory analysis of the primary endpoints

The same statistical model as used for the primary analysis (Sections 7.3.1 of the CTP) will be repeated for the primary endpoints but with all sources of variation ("sequence", "subjects within sequences", "period", "treatment") considered as fixed effects.

Primary PK endpoints will be assessed descriptively. The analysis of standard PK parameters is performed according to BI standards (4).

### 7.5 SECONDARY ENDPOINTS

### 7.5.1 Key secondary endpoints

This section is not applicable as no key secondary endpoint has been specified in the protocol.

### 7.5.2 Secondary endpoints

The secondary endpoints will be statistically analysed in the same way as for the primary endpoints. The endpoints will also be assessed descriptively. The analysis of standard PK parameters is performed according to BI standards (4).

See <u>Section 7.4</u> of this TSAP for details regarding exclusion of PK parameters and plasma concentrations.

### 7.7 EXTENT OF EXPOSURE

Descriptive statistics are planned for this section of the report, by treatment and overall.

### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

### 7.8.1 Adverse Events

AEs will be coded with the most recent version of MedDRA.

The analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and not on the number of AEs.

For analysis, multiple AE occurrence data on the eCRF will be collapsed into one event provided that all of the following applies:

- All AE attributes are identical (lower level term, intensity, action taken, therapy required, seriousness, reason for seriousness, relationship, outcome, AESI)
- The occurrences were time-overlapping or time-adjacent (time-adjacency of two occurrences is given if the second occurrence started at most 1 hour after the first occurrence ended)

For further details on summarization of AE data, please refer to "Analysis and Presentation of Adverse Event Data from Clinical Trials" (7) and "Handling of missing and incomplete AE dates" (3).

The analysis of AEs will be based on the concept of treatment emergent AEs. That means that all AEs will be assigned to screening or on-treatment phases as defined in Section 6.1. AEs will be analysed based on actual treatments, as defined in Table 6.1: 2.

An overall summary of AEs will be presented. This overall summary will comprise summary statistics for the class of other significant AEs according to ICH E3 (8) and for the class of AESIs.

**CTP:** The following are considered as AESIs:

- *Hepatic injury* 
  - A hepatic injury is defined by the following alterations of hepatic laboratory parameters:
  - $\circ$  An elevation of AST (aspartate transaminase) and/or ALT (alanine transaminase)  $\geq$ 3-fold ULN combined with an elevation of total bilirubin  $\geq$ 2-fold ULN measured in the same blood sample, or
  - $\circ$  Aminotransferase (ALT, and/or AST) elevations  $\geq$ 10 fold ULN

The investigator had to classify on the eCRF whether an observed AE was an AESI or not.

According to ICH E3 (8) AEs classified as "other significant" need to be reported and will include those non-serious and non-significant AEs

- (i) which are marked haematological or other lab abnormalities, or
- (ii) which were reported with "action taken = discontinuation" or "action taken = reduced", or
- (iii) which lead to significant concomitant therapy as identified by the Clinical Monitor/Investigator at a Medical Quality Review Meeting.

The frequency of subjects with AEs will be summarised by treatment, primary SOC and preferred term. AEs which were considered by the investigator to be drug related will be summarised separately. Separate tables will also be provided for subjects with SAEs, subjects with AESIs and subjects with other significant AEs (according to ICH E3 (8)). The frequency of subjects with AEs and the frequency of subjects with AEs considered by the investigator to be drug related will also be summarised by maximum intensity, primary SOC and preferred term.

The SOCs and preferred terms within SOCs will be sorted by descending frequency over all treatment groups.

For disclosure of AE data on ClinicalTrials.gov, the frequency of subjects with non-serious AEs occurring with an incidence of greater than 5 % (in preferred terms) will be summarised by treatment, primary SOC and preferred term. The frequency of subjects with SAEs will also be summarised.

For disclosure of AE data in the EudraCT register, the frequency of AEs, the frequency of non-serious AEs with an incidence of greater than 5 % (in preferred terms) and the frequency of SAEs will be summarized.

For support of lay summaries, the frequency of subjects with drug-related SAEs will be summarized by treatment, primary SOC and preferred term.

If the subject reports headaches during the treatment period further information about the duration of headache, location, characteristics, and signs and symptoms were recorded. The information will be summarized with descriptive statistics.

### 7.8.2 Laboratory data

TSAP for BI Trial No: 1402-0010

The analyses of laboratory data will be descriptive in nature and will be based on BI standards "Display and Analysis of Laboratory Data" (9).

Analyses will be based on normalised values, which means transforming to a standard unit and a standard reference range. The original values will be analysed if the transformation into standard unit is not possible for a parameter.

Descriptive statistics of laboratory values over time and for the difference from baseline (see Section 6.7) will be provided. Frequency tables of changes between baseline and last value on treatment with respect to the reference range will be presented.

Possibly clinically significant abnormal laboratory values are only those identified either in the Investigator's comments or at the Report Planning Meeting at the latest. It is the Investigator's responsibility to decide whether a lab value is clinically significant abnormal or not. Standard or project-specific rules for flagging clinically significant values in an automated manner will not be applied in this study.

Clinically relevant findings in laboratory data will be reported as baseline conditions (prior to first administration of study treatment) or as AEs (after first administration of study treatment) if judged clinically relevant by the investigator, and will be analyzed as such.

# 7.8.3 Vital signs

The analyses of vital signs (blood pressure and pulse rate) will be descriptive in nature. Descriptive statistics of vital signs over time (baseline and on-treatment measurements, cf. Table 6.1: 2, only) and for the difference from baseline (see Section 6.7) will be provided.

Clinically relevant findings in vital signs data will be reported as baseline conditions (prior to first administration of study treatment) or as AEs (after first administration of study treatment) if judged clinically relevant by the investigator, and will be analyzed as such.

### 7.8.4 ECG

Relevant ECG findings will be reported as relevant medical history/baseline condition (if a condition already exists before first administration of study treatment) or as AE (if condition emerges after first administration of study treatment) and will be summarized as such. No separate listing or analysis of ECG findings will be prepared.

### **7.8.5** Others

Physical examination findings will be reported as relevant medical history/baseline condition (if a condition already exists before first administration of study treatment) or as AE (if condition emerges after first administration of study treatment) and will be summarized as such. No separate listing or analysis of physical examination findings will be prepared.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Reports of C-SSRS will be reported as AEs as described in CTP Section 5.2.6.1.7 and will be summarized as such. Results of the C-SSRS will only be listed. No further analysis will be prepared.

Clinically relevant findings of the neurological examination will be reported as relevant medical history/baseline condition (if a condition already exists before first administration of study treatment) or as AE (if condition emerges after first administration of study treatment) and will be summarized as such. No separate listing or analysis of neurological examinations will be prepared.

### **REFERENCES** 8.

| 1 | CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9; Note For Guidance on Design, Conduct, Analysis and Evaluation of Clinical Trialss, current version |
|---|---|
| 2 | 001-MCS-40-413_1.0: "Identify and Manage Important Protocol Deviations (iPD)", current version; IDEA for CON |
| 3 | KM Asset BI-KMED-BDS-HTG-0035: "Handling of missing and incomplete AE dates", current version; KMED |
| 4 | 001-MCS-36-472_RD-01: "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies", current version; IDEA for CON |
| 5 | KM Asset BI-KMED-BDS-HTG-0045: "Reporting of Clinical Trials and Project Summaries", current version; KMED |
| 6 | 001-MCS-36-472_RD-03: "Description of Analytical Transfer Files and PK/PD Data Files", current version; IDEA for CON |
| 7 | KM Asset BI-KMED-BDS-HTG-0041: "Analysis and Presentation of Adverse Event Data from Clinical Trials", current version; KMED |
| 8 | CPMP/ICH/137/95: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version |
| 9 | KM Asset BI-KMED-BDS-HTG-0042: "Display and Analysis of Laboratory Data", current version; KMED |

TSAP for BI Trial No: 1402-0010 
Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1402-0010 

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

### **10. HISTORY TABLE**

Table 10: 1 History table

| Version | Date<br>(DD-MMM-YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Final | 06-AUG-2019 | | None | This is the final TSAP |